CLINICAL TRIAL: NCT05499286
Title: A Mindfulness-Based Intervention to Improve CPAP Adherence in Adolescents With Obstructive Sleep Apnea
Brief Title: A Mindfulness-Based Intervention to Improve CPAP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Indra Narang, Principal Investigator, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1000068799
Record Dates: First submitted 2022-04-25; First posted 2022-08-12 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Obstructive Sleep Apnea (Moderate to Severe); Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindfulness Program (Active Comparator): Participants will attend an online mindfulness program known as the Mindful Awareness and Resilience Skills for Adolescents (MARS-A) program.
  Interventions: Other: Mindfulness Program
- Online Peer Support Program (No Intervention): Participants will attend an online peer support program where they will engage with each other by sharing experiences while providing advice and emotional support.

INTERVENTIONS:
Other: Mindfulness Program — Mindful Awareness and Resilience Skills for Adolescents (MARS-A) Curriculum
  Arms: Mindfulness Program

SUMMARY:
The main purpose of this study is to assess the effectiveness of a mindfulness-based intervention in improving CPAP use compared to online peer support

ELIGIBILITY:
Inclusion Criteria:

* Adolescent age (13-18 years)
* Confirmed diagnosis of moderate or severe OSA
* Adolescent should have the capacity to consent themselves

Exclusion Criteria:

* Known developmental delay such that they are not able to participate in the study;
* Neuromuscular disorders
* Central sleep apnea
* Known diagnosis of severe psychiatric illnesses (e.g. suicidal ideation)
* Limited knowledge and proficiency in English to complete the study as judged by the clinical team

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 102 (Estimated)
Dates: Start 2020-06-28 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
The effectiveness of MBI for CPAP adherence. | Week 4-12
  The primary objective is to evaluate the effectiveness of a mindfulness-based intervention (MBI) in improving CPAP adherence in adolescents with OSA when compared to online peer support. Adherence to CPAP will be measured objectively as hours of usage of CPAP per night.

SECONDARY OUTCOMES:
The effects of increased adherence on mental, physical, and psychosocial statuses. | Week 4-12
  Evaluate the effects of increased CPAP adherence on daytime sleepiness, HRQOL, psychosocial functioning and mental health status (e.g. anxiety and depression). This will be measured by administering questionnaires at baseline, before intervention, after intervention and again at follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Indra Narang, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No